CLINICAL TRIAL: NCT02126124
Title: A Prospective, Double Blind, Randomized, Controlled Study to Evaluate the Safety and Efficacy of the Deep Transcranial Magnetic Stimulation (DTMS) (With the H-ADD Coil) Intended as an Aid to Smoking Cessation.
Brief Title: Evaluation of Deep Transcranial Magnetic Stimulation (DTMS) With the H-ADD Coil as an Aid to Smoking Cessation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BR-SMOK-01
Record Dates: First submitted 2014-04-27; First posted 2014-04-29 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2019-11

CONDITIONS: Smoking Cessation
Keywords: Brainsway, dTMS, Deep Transcranial Magnetic Stimulation, Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active dTMS Treatment (Active Comparator): Brainsway Deep TMS Treatment
  Interventions: Device: Active dTMS Treatment
- Sham Treatment (Sham Comparator): Brainsway Sham Treatment
  Interventions: Device: Sham Treatment

INTERVENTIONS:
Device: Sham Treatment — In the sham treatment, the electrical field induced by the sham coil cannot invoke any action potentials and if no action potentials are induced, then the electric field is insignificant and there is no treatment effect on the the brain.
  Other Names: Brainsway Sham Treatment
  Arms: Sham Treatment
Device: Active dTMS Treatment — Deep Transcranial Magnetic Stimulation (dTMS) is a new form of TMS which allows direct stimulation of deeper neuronal pathways than the standard TMS. The Brainsway Coil is a novel dTMS coil desigend to allow deeper brain stimulation without significant increase of electric fields induced in superficial cortical regions.
  Other Names: Brainsway Deep TMS Treatment
  Arms: Active dTMS Treatment

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of DTMS compared to sham treatment as an aid to smoking cessation in chronic, heavy (>10 cigarettes/day) cigarette smokers.

DETAILED DESCRIPTION:
This is a multi center, randomized, double blind study to evaluate the safety and effectiveness of the device as an aid to smoking cessation. Treatment will be administered over a 6 week period and follow-up assessments will be conducted at 4 months. The clinical study design includes multiple measurements of safety and effectiveness parameters. The design is meant to demonstrate that the device shows superiority compared to sham treatment over six treatment weeks, at the 4 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 22-70 years old.
* Chronic, heavy (>10 cigarettes/day) smokers, who smoke for more than 1 year, with no period of abstinence for greater than 3 months during the past year.
* Subjects who are motivated to quit smoking (with responses "very likely," or "somewhat likely" to the motivation questionnaire).
* Satisfactory answers on safety screening questionnaire for transcranial magnetic stimulation (Keel 2001).
* Gave informed consent for participation in the study.

Exclusion Criteria:

* Currently on Nicotine Replacement Therapy (NRT) or smoking cessation drugs (e.g., Zyban, Chantix, etc.) or undergoing behavioral smoking cessation interventions
* Cognitive or functional disability, diagnosed according to DSM-IV-TR criteria.
* Active psychiatric disorder according to DSM IV (Axis I and Axis II) criteria within the last year.
* Current alcohol or other substance abuse or dependence.
* Alcohol or other substance abuse or dependence during the last 12 months before recruitment.
* Subject is smoking any other form of tobacco or other substances.
* Subject is taking psychotropic medications on a regular basis.
* Subjects with a high risk for severe violence or suicidality as assessed during the screening interview.
* Subjects who suffer from an unstable physical disease such as high blood pressure (>150 mmHg systolic / diastolic > 110 mmHg) or acute, unstable cardiac disease.
* History of epilepsy or seizure (EXCEPT those therapeutically induced by ECT).
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or history of significant head injury or trauma with loss of consciousness for > 5 minutes.
* History of any metal in the head (outside the mouth).
* Metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or implanted medical pumps.
* Individuals with a significant neurological disorder or insult including, but not limited to:

  * Any condition likely to be associated with increased intracranial pressure
  * Space occupying brain lesion
  * History of cerebrovascular accident
  * Transient ischemic attack within two years
  * Cerebral aneurysm
  * Dementia
  * Mini Mental State Exam score of less than or equal to 24
  * Parkinson's disease
  * Huntington's chorea
  * Multiple sclerosis
* Subjects suffering from frequent and severe migraine headaches.
* Subjects suffering from significant hearing loss.
* Subjects taking pro-convulsant medications (e.g., antidepressants or antipsychotic medications).
* Previous treatment with TMS.
* Subjects who cannot communicate reliably with the investigator or who are not likely to cope with the requirements of the experiment.
* Participation in a clinical trial within the last 30 days before the beginning of this clinical trial or similar participation in another clinical trial.
* Known or suspected pregnancy or lactation.
* Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2014-08-20 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Continuous Quit Rate | 4 week
  The primary objective is to compare the four-week continuous quit rate (CQR), representing abstinence during a consecutive 4 week period during the treatment phase, between the two treatment groups.

SECONDARY OUTCOMES:
Number of Cigarettes Smoked Per Day | 4 Weeks
  The secondary objective is to compare number of cigarettes smoked per day (per diary data) for all subjects.

OTHER OUTCOMES:
Long term CQR | 4 Months
  Long-term continuous quit rates (CQR) at four months.
Withdrawal Symptoms | 6 Weeks
  Effect on withdrawal symptoms as measured by weekly scales measuring nicotine craving and dependence/withdrawal, including Fagerstrom Test for Nicotine Dependence (FTND), Minnesota Nicotine Withdrawal Scale Self-Report (MNWS), Tobacco Craving Questionnaire-Short Form (TCQ-SF) and Nicotine Craving Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mark George, MD, Principal Investigator — Medical University of South Carolina; Abraham Zangen, PhD, Principal Investigator — Soroka University Medical Center; Kathleen Brady, MD., PhD, Principal Investigator — Medical University of South Carolina
Locations (18):
- United States (14):
  - Pacific Institute of Medical Research, Los Angeles, California
  - University of California - San Diego Medical Center, San Diego, California
  - TMS Center of Colorado, Denver, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - Advanced Mental Health Care Inc. - Juno Beach, Juno Beach, Florida
  - Advanced Mental Health Care Inc. - Royal Palm Beach, Royal Palm Beach, Florida
  - McLean Hospital - TMS Services, Belmont, Massachusetts
  - Premier Psychiatric Group, Lincoln, Nebraska
  - Premier Psychiatric Group, Omaha, Nebraska
  - Mount Sinai Hospital, New York, New York
  - Columbia University / New York State Psychiatric Institute, New York, New York
  - Lindner Center of HOPE, University of Cinicnnati College of Medicine, Cincinnati, Ohio
  - Medical University Of South Carolina (MUSC), Charleston, South Carolina
  - Senior Adults Specialty Research, Austin, Texas
- Center for Addiction and Mental Health (CAMH), Toronto, Ontario, Canada
- Israel (3):
  - Beer Yaacov Mental Health Center, Beer Yaacov
  - Soroka Medical Center, Beersheba
  - Lev Hasharon, Netanya

REFERENCES:
- [Derived] Zangen A, Moshe H, Martinez D, Barnea-Ygael N, Vapnik T, Bystritsky A, Duffy W, Toder D, Casuto L, Grosz ML, Nunes EV, Ward H, Tendler A, Feifel D, Morales O, Roth Y, Iosifescu DV, Winston J, Wirecki T, Stein A, Deutsch F, Li X, George MS. Repetitive transcranial magnetic stimulation for smoking cessation: a pivotal multicenter double-blind randomized controlled trial. World Psychiatry. 2021 Oct;20(3):397-404. doi: 10.1002/wps.20905. PMID 34505368